CLINICAL TRIAL: NCT03404882
Title: Enhancing Peer-support Experience for Patients Discharged From Acute Psychiatric Care: Protocol for a Randomized Controlled Pilot Trial
Brief Title: Peer Support Experience for Patients Discharged From Acute Psychiatric Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00078427
Record Dates: First submitted 2018-01-08; First posted 2018-01-19 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Depression; Bipolar Disorder; Schizophrenia
MeSH Terms: conditions — Depression; Bipolar Disorder; Schizophrenia | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This will be a longitudinal, prospective, parallel design, three arm, rater-blinded randomized clinical trial with a recruitment period of six months and an observation period of 12 months for each participant.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to treatment group allocation by not involving them in discussions about study participants and not granting them access to the database which contains the randomization code. In addition, study participants will be asked not to reveal their treatment allocation to their assessor. Moreover, these assessors will not be involved in data analysis. To test the success of blinding we will ask the assessor to guess the treatment group for each participant at six and 12-month follow-up. After data collection is complete all data will undergo a blind review for the purposes of finalizing the planned analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- text messaging plus peer support arm (Experimental): Patients will be assigned a peer support worker who will visit them during the last week of their inpatient stay to introduce themselves and build rapport before patients are discharged into the community. The peer support workers will visit the participants up to eight times over a six month period. The peer support workers will offer the opportunity for interactive text message support for six months. In addition to peer support, participants in this arm of the study will receive daily supportive text messages from an automated online application and reminder text messages for their community clinic/program appointments.
  Interventions: Behavioral: Supportive/reminder text messaging plus peer support
- supportive/reminder text message only arm (Active Comparator): Patients in the supportive/reminder text message only arm of the study will receive daily supportive text messages from the automated online application and reminder text messages for their community clinic/program appointments.
  Interventions: Behavioral: Supportive/reminder text messaging
- Control arm (No Intervention): Patients in the control arm of the study will receive the usual follow-up appointment offered to all patients who are discharged from acute care. However, they will not receive peer support or supportive/reminder text messages.
- peer support only arm (Active Comparator): Patients will be assigned a peer support worker who will visit them during the last week of their inpatient stay to introduce themselves and build rapport before patients are discharged into the community. The peer support workers will visit the participants up to eight times over a six month period. The peer support workers will offer the opportunity for interactive text message support for six months. Patients will not receive daily supportive/reminder text messages
  Interventions: Behavioral: Peer support only

INTERVENTIONS:
Behavioral: Supportive/reminder text messaging plus peer support — Regular supportive/reminder text message will be delivered to patients who will also receive face to face and interactive text message support from peer support workers
  Arms: text messaging plus peer support arm
Behavioral: Supportive/reminder text messaging — Regular supportive/reminder text message will be delivered to patients who will NOT receive any face to face or interactive text message support from peer support workers
  Arms: supportive/reminder text message only arm
Behavioral: Peer support only — face to face support from peer support workers but no interactive or daily supportive/reminder text messages
  Arms: peer support only arm

SUMMARY:
The aim of the project is to conduct a four arm randomized controlled pilot trial to evaluate the effectiveness of an innovative peer support program that incorporates leadership training, mentorship, recognition, reward systems and supportive/reminder text messaging for patients discharged from acute (hospital) care. Methods and analysis: This is a prospective, rater-blinded, four arm randomized controlled trial. 180 patients discharged from acute psychiatric care in Edmonton, Alberta, Canada will be randomized to one of four conditions: treatment as usual follow-up care, enrollment in usual follow-up care plus daily supportive/reminder text messages, enrollment in a peer support system plus daily supportive/reminder text messages or enrollment in a peer support system without daily supportive text messages. Patients in each group will complete evaluation measures (e.g., recovery, general symptomatology, functional outcomes) at baseline, six and twelve weeks & six and 12 months. Service utilization data and data regarding the experience of the peer support workers will also be collected. Data will be analyzed with descriptive statistics, repeated measures, and correlational analyses. We hypothesize that patients enrolled in the peer support system plus daily supportive/reminder text messages condition will achieve superior outcomes in comparison to other groups. Peer support worker experience will be derived from exploratory data analysis.

DETAILED DESCRIPTION:
Background and Rationale Peer support is emotional, social and practical help provided by non-professionals to assist people with sustaining health behaviours. The peer support workers share a similar condition as patients, effectively manage their condition, and have received training to provide support. Peer support is provided to people with psychological health complaints by peer supporter workers with lived experience, and the position of peer support worker may include activities such as advocacy, connecting patients with resources, and experiential sharing, among others .

Peer support is consistent with the recovery paradigm in mental health, and is differentiated from psychiatric models of traditional diagnosis and treatment. The purported mechanisms through which peer support may function are through experiential knowledge sharing, modeling of adaptive coping strategies, social comparison, and enhancing social support. Moreover, peer support may be particularly useful for clients who have difficulty engaging in conventional services . It may be the case that peer support systems can serve as an entry point into the healthcare system for 'hardly reached' individuals and at the very least, serve as a means of providing supportive services for those who would otherwise not engage in treatment. In addition, providing peer support may offer benefits to the peer supporter her/himself, by enhancing feelings of competence and personal value .

Peer support is valued in recovery-oriented models of mental health and is becoming increasingly implemented organizationally [see Myrick and del Vecchio for a discussion]. Many studies have reported positive effects of peer support, including lower inpatient service use, better relationships with providers, and increased engagement. However, a recent rigorous evaluation of randomized controlled trials (RCTs) of peer support studies reported that outcomes were generally mixed and often non-significant. In their review, the authors noted a high degree of bias and methodological limitations in the studies they reviewed, and concluded that "peer support programmes should be implemented within the context of high quality research projects wherever possible".

In addition to methodological improvements of research on peer support, there is a need to further develop the peer support workforce. Identified areas of development for peer support programs include: how to define "peerness", role clarity and integration with existing systems, credentialing, and workforce development. Within our local context, in the province of Alberta, Canada, peer support for patients has been in existence for many years. Anecdotal evidence suggests there is low uptake and high attrition for peer support worker roles within the province. There has been a drive to develop curricula and organizational infrastructure to formally train and support peer support workers. Administrators who have worked with peer support workers suggest the lack of adequate incentives may contribute to peer support workforce challenges. Relatedly, there are often limited incentives for mental health professionals to provide supervision and mentorship for peer support workers locally.

In summary, the existing literature suggests there is opportunity for innovation in peer support programs, and there is a need for rigorous methodology to better evaluate outcomes from peer support programs. There is also a need to further develop the peer support workforce. The current paper describes a randomized controlled trial that is designed to systematically evaluate a novel peer support model termed the "Edmonton Peer Support System" (EPSS), which incorporates innovative features of service delivery (i.e., an incentive-based model of training, text messaging) and rigorous methodological design to minimize bias and confounds (e.g., comprehensive measures of outcome; methodological design features including longitudinal, prospective, three arm parallel design, and rater-blinding).

One of the innovative features of this study is the incorporation of text messaging. Text messaging is a relatively low cost, high impact, and easily scalable program that uses existing technology, is devoid of geographic barriers, and is easily accessible to end users. There is evidence that supportive text messaging demonstrates positive effects in terms of symptom improvement and patient satisfaction. For example, patients with depression and comorbid alcohol use disorder showed significantly lower depressive symptoms on standardized self-report than a similar patient group who did not receive messages [large effect size)(9)]. A second randomized trial demonstrated similar results [(Cohen's d= 0.67)(10)]. In terms of satisfaction, over 80% of subscribers reported that a texting program improved their mental health.

There is also evidence that reminder text messaging improves appointment attendance rates. For example, in a systematic review and meta-analysis of eight randomized controlled trials involving 6615 participants, the authors found moderate quality evidence from seven studies (5841 participants) that mobile text message reminders improved the rate of attendance at healthcare appointments compared to no reminders [risk ratio (RR) 1.14 (95% confidence interval (CI) 1.03 to 1.26)]. They also found that text messaging reminders were similar to telephone reminders in terms of their effect on attendance rates, yet cost less than telephone reminders.

Another innovative feature of this study is the incorporation of a peer support incentive system. As discussed, the peer support workforce has been identified as an area in need of development, including role clarity, integration with healthcare professionals, and credentialing. Specifically, a lack of a "career ladder" or a clear movement within positions of peer support work has been identified, with movement possible laterally (but not upward) within many program structures. In this project, peer support workers will participate in an incentive based system that formally recognizes performance. The EPSS is structured as follows:

* Peer support workers are people with lived mental health experience who are at a point in their personal recovery where they consistently demonstrate the ability to share their individual story in a manner that inspires hope and builds relationships with others. Peer support workers who are employed by Alberta Health Services (AHS), our provincial health authority, will be invited to enroll as foundational members of the EPSS.
* Members will be provided with formalized training developed within our health region, involving knowledge training, practice, and ongoing meetings throughout offering the program to assist peer support workers in adhering to principles consistent with a peer support framework and recovery philosophy and problem-solving concerns or challenges that may arise. Peer support workers will receive clinical support/mentorship from mental health therapists.
* Patient beneficiaries of EPSS will receive supportive face-to-face visits, phone calls, and interactive text message support from their peer support workers. They will also receive reminder text messages for their appointments.
* Patient beneficiaries will be enrolled as associate members of the EPSS and will be provided with training to act as peer support workers when they are an advanced stage in their recovery. At this time they can apply for AHS peer support worker roles as available.
* Contributions of peer support workers will be recognized via attainment of different levels of membership (e.g. "star" levels) and certificates of recognition (bearing logos of collaborating institutions) at formal ceremonies. Star-level recognition will be categorized into: Silver Star Memberships (five stars), Gold Star Memberships (ten stars), and Star Fellowships (twenty stars).
* Contributions of mental health therapists towards supporting/mentoring peer support workers will also be recognized through star memberships and certificates at formal ceremonies.

The hope of EPSS is to increase compassion and decrease stigma, foster multi-disciplinary teamwork, incorporate client/caregiver experiences, and strengthen service provider skills and abilities. Our proposed EPSS will provide training for those with mental health challenges that will enable them to contribute providing compassionate care for mental health patients. This program philosophy is aligned with regional goals relating to improvement of mental health services in our province.

Aim and Objectives The aim of the project is to evaluate the effectiveness of an EPSS which incorporates leadership training, mentorship, recognition, reward systems and supportive/reminder text messaging for patients discharged from acute (hospital) care. The client outcomes will be organized according to: recovery variables (e.g., recovery, stigma), functional variables (quality of life, employment), symptom variables (psychological symptoms, general outcomes), and service variables (e.g., heath service utilization, cost, satisfaction), as further described in Methods and Analysis. Peer support worker outcomes will also be evaluated, including effectiveness, job satisfaction, acceptability, and recovery.

The objectives of the project include:

1. To compare mean changes in recovery, functional outcomes, clinical symptoms, and service variables after six weeks, twelve weeks, six months and twelve months for patients in each of the three arms: those discharged from acute care and enrolled in peer support system plus daily supportive/reminder text messages; those with usual follow-up care plus daily supportive/reminder text messages, and those receiving usual follow-up care.
2. To assess job satisfaction, acceptability, and recovery of peer support workers at six and twelve months.
3. To assess job satisfaction among mental health therapists offering support and mentorship for peer support workers.

Hypothesis The investigators hypothesize that patients enrolled in the peer support system plus daily supportive/reminder text messages will achieve superior outcomes compared to patients enrolled in the other arms of the study on each outcome measure used. In turn, patients enrolled in peer support will have superior outcomes to patients enrolled in the treatment as usual condition.

Data Analysis:

Initially, we aimed to deploy intention-to-treat analysis, whereby patient data are analyzed according to their original assigned groups, regardless of time spent in the study. However, after randomization and due to clinical logistic reasons, a significant number of patients did not receive access to the Peer Support Worker service in the two intervention arms of Peer Support Worker. Thus we have made a strategic decision to adapt the protocol to a Controlled Observational Study and to change the analysis approach to as-treated, rather than intention-to-treat to maximize the investigational value of the study without compromising or biasing outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18-65 years of age, able to provide informed written consent, have been diagnosed with an enduring mental health condition and are ready for discharge from an acute care facility within the Edmonton Zone with community mental health follow-up.
* Patients should have a mobile handset capable of receiving text messages. Mobile phone handsets and top-up call credit of up to 10 dollars monthly will be provided to those who satisfy the inclusion criteria but do not have mobile phones.

Exclusion Criteria:

* Patients will be ineligible if they do not meet the above inclusion criteria, if they have only an addictive disorder but no mental health diagnosis, are not capable of reading text messages from a mobile device, or will be out of town during the 12 month follow-up period.
* Patients are also ineligible if they do not consent to take part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Core Outcome Measure | 6 & 12 Weeks and 6 $ 12 Months
  Core outcome measure has 34 question measure covering 5 sub-scales
  * Relation to self and others
  * Daily living and role functioning
  * Depression and anxiety
  * Impulsive and addictive behaviour
  * Psychosis
  Sub-scale and overall mean scores also range from 0 to 4. Four of the five subscale scores and the BASIS-32 average are computed by averaging the ratings for component items using the number of non-missing items as the denominator. The score range from 0 to 128
Changes in Health of Nations Outcome Scale (HoNOS) score from Baseline | 6 & 12 Weeks and 6 $ 12 Months
  HoNOS measures the symptom severity and social functioning across time. It has 12 items that measure behaviour, impairment, symptoms and social functioning. The items are rated on a scale of 0-4 and the results or changes in ratings are known as outcomes and may be attributed to services provided. The scores range from 0 to 48.

SECONDARY OUTCOMES:
Perceived Discrimination Scale score | 6 & 12 Weeks and 6 & 12 Months
  This is a 5 scale item with each scale scored either from 0-3, 0-4 or 0-6, with 38 questions. The score ranges from 0 to 145 with calculation of each scale mean, standard deviation and alpha for each patient.
World Health Organization Quality of Life Brief instrument (WHOQOL-BREF) score | 6 & 12 Weeks and 6 $ 12 Months
  The WHOQOL-BREF produces a quality of life profile. It is possible to derive four domain scores. The mean score of items within each domain is used to calculate the domain score. Mean scores are then multiplied by 4 in order to make domain scores comparable with the scores used in the WHOQOL-100. Raw scores are then transformed to scores which range from 0-100 scale.
Patient Satisfaction/Experience Questionnaire | 6 & 12 Months
  This scale has 10 questions with a Liket scale with five options for each question. The score range from 10 to 50
Rates of Health services utilization | 6 & 12 Months
  Rates of use, inpatient admissions and length of stay, readmissions, completed appointments, Emergency Department presentations, Emergency Medical Services use, community services appointments, crisis and urgent service calls, no show rates.
Cost of Health services utilized | 6 & 12 Months
  Cost of use, inpatient admissions and length of stay, re-admissions, completed appointments, Emergency Department presentations, Emergency Medical Services use, community services appointments, crisis and urgent service calls, and no show cost.
Peer Support Worker Effectiveness | 6 & 12 Months
  Will be assessed through qualitative interviews of key informants and focus group discussions
Peer Support Worker Job satisfaction | 6 & 12 Months
  Will be assessed through qualitative interviews of key informants and focus group discussions
Peer Support Worker Acceptability | 6 & 12 Months
  Will be assessed through qualitative interviews of key informants and focus group discussions
Recovery Assessment Scale score for Peer Support workers | 6 & 12 Months
  The Recovery Assessment Scale has 24 items. It is a Likert scale with 5 rating categories.
  "completely true" which are scored 1, 2, 3 and 4 respectively giving a range of scores from 38 to 152.
Recovery Assessment Scale score | 6 & 12 Weeks and 6 &12 Months
  The Recovery Assessment Scale has 24 items. It is a Likert scale with 5 rating categories for consumers to select from: "untrue"; "a bit true"; "mostly true" and "completely true" which are scored 1, 2, 3 and 4 respectively giving a range of scores from 38 to 152.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Royal Alex Hospital, Edmonton, Alberta
  - Alberta Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Proudfoot JG, Jayawant A, Whitton AE, Parker G, Manicavasagar V, Smith M, Nicholas J. Mechanisms underpinning effective peer support: a qualitative analysis of interactions between expert peers and patients newly-diagnosed with bipolar disorder. BMC Psychiatry. 2012 Nov 9;12:196. doi: 10.1186/1471-244X-12-196. PMID 23140497
- [Background] Jacobson N, Trojanowski L, Dewa CS. What do peer support workers do? A job description. BMC Health Serv Res. 2012 Jul 19;12:205. doi: 10.1186/1472-6963-12-205. PMID 22812608
- [Background] Onken SJ, Craig CM, Ridgway P, Ralph RO, Cook JA. An analysis of the definitions and elements of recovery: a review of the literature. Psychiatr Rehabil J. 2007 Summer;31(1):9-22. doi: 10.2975/31.1.2007.9.22. PMID 17694711
- [Background] Myrick K, Del Vecchio P. Peer support services in the behavioral healthcare workforce: State of the field. Psychiatr Rehabil J. 2016 Sep;39(3):197-203. doi: 10.1037/prj0000188. Epub 2016 May 16. PMID 27183186
- [Background] Chinman M, George P, Dougherty RH, Daniels AS, Ghose SS, Swift A, Delphin-Rittmon ME. Peer support services for individuals with serious mental illnesses: assessing the evidence. Psychiatr Serv. 2014 Apr 1;65(4):429-41. doi: 10.1176/appi.ps.201300244. PMID 24549400
- [Background] Lloyd-Evans B, Mayo-Wilson E, Harrison B, Istead H, Brown E, Pilling S, Johnson S, Kendall T. A systematic review and meta-analysis of randomised controlled trials of peer support for people with severe mental illness. BMC Psychiatry. 2014 Feb 14;14:39. doi: 10.1186/1471-244X-14-39. PMID 24528545
- [Background] Silver J, Nemec PB. The role of the peer specialists: Unanswered questions. Psychiatr Rehabil J. 2016 Sep;39(3):289-91. doi: 10.1037/prj0000216. PMID 27618464
- [Background] Agyapong VI, Ahern S, McLoughlin DM, Farren CK. Supportive text messaging for depression and comorbid alcohol use disorder: single-blind randomised trial. J Affect Disord. 2012 Dec 10;141(2-3):168-76. doi: 10.1016/j.jad.2012.02.040. Epub 2012 Mar 29. PMID 22464008
- [Background] Agyapong VIO, Juhas M, Ohinmaa A, Omeje J, Mrklas K, Suen VYM, Dursun SM, Greenshaw AJ. Randomized controlled pilot trial of supportive text messages for patients with depression. BMC Psychiatry. 2017 Aug 2;17(1):286. doi: 10.1186/s12888-017-1448-2. PMID 28768493
- [Background] Agyapong VI, McLoughlin DM, Farren CK. Six-months outcomes of a randomised trial of supportive text messaging for depression and comorbid alcohol use disorder. J Affect Disord. 2013 Oct;151(1):100-4. doi: 10.1016/j.jad.2013.05.058. Epub 2013 Jun 22. PMID 23800443
- [Background] Agyapong VI, Mrklas K, Juhas M, Omeje J, Ohinmaa A, Dursun SM, Greenshaw AJ. Cross-sectional survey evaluating Text4Mood: mobile health program to reduce psychological treatment gap in mental healthcare in Alberta through daily supportive text messages. BMC Psychiatry. 2016 Nov 8;16(1):378. doi: 10.1186/s12888-016-1104-2. PMID 27821096
- [Background] Gurol-Urganci I, de Jongh T, Vodopivec-Jamsek V, Atun R, Car J. Mobile phone messaging reminders for attendance at healthcare appointments. Cochrane Database Syst Rev. 2013 Dec 5;2013(12):CD007458. doi: 10.1002/14651858.CD007458.pub3. PMID 24310741
- [Background] Alberta AH-G of. Valuing mental health: Next steps: Alberta Health website [Internet]. [cited 2018 Jan 3]. Available from: http://www.health.alberta.ca/initiatives/Mental-Health-Review.html
- [Background] Edmonton C of. 2016 Municipal Census Results [Internet]. 2017 [cited 2017 Sep 14]. Available from: https://www.edmonton.ca/city_government/facts_figures/municipal-census-results.aspx
- [Background] Giffort D, Schmook A, Woody C, Vollendorf C, Gervain M. Recovery Assessment Scale. Cambridge, MA: Human Services Research Institute; 1995
- [Background] Major B, O'Brien LT. The social psychology of stigma. Annu Rev Psychol. 2005;56:393-421. doi: 10.1146/annurev.psych.56.091103.070137. PMID 15709941
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] What is HoNOS? [Internet]. [cited 2018 Jan 4]. Available from: http://www.rcpsych.ac.uk/traininpsychiatry/conferencestraining/resources/honos/whatishonos.aspx
- [Background] Eisen SV, Normand SL, Belanger AJ, Spiro A 3rd, Esch D. The Revised Behavior and Symptom Identification Scale (BASIS-R): reliability and validity. Med Care. 2004 Dec;42(12):1230-41. doi: 10.1097/00005650-200412000-00010. PMID 15550803
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Guidelines for Good Clinical Practice (GCP) for Trials on Pharmaceutical Products. WHO Technical Report Series, No. 850, Annex 3 - WHO Expert Committee on Selection and Use of Essential Medicines, Sixth Report, 1993 [Internet]. [cited 2017 Nov 22]. Available from: http://apps.who.int/medicinedocs/en/d/Jwhozip13e/
- [Result] Sokol R, Fisher E. Peer Support for the Hardly Reached: A Systematic Review. Am J Public Health. 2016 Jul;106(7):e1-8. doi: 10.2105/AJPH.2016.303180. Epub 2016 May 19. PMID 27196645
- [Derived] Shalaby R, Vuong W, Eboreime E, Surood S, Greenshaw AJ, Agyapong VIO. Patients' Expectations and Experiences With a Mental Health-Focused Supportive Text Messaging Program: Mixed Methods Evaluation. JMIR Form Res. 2022 Jan 11;6(1):e33438. doi: 10.2196/33438. PMID 35014972
- [Derived] Urichuk L, Hrabok M, Hay K, Spurvey P, Sosdjan D, Knox M, Fu A, Surood S, Brown R, Coulombe J, Kelland J, Rittenbach K, Snaterse M, Abba-Aji A, Li XM, Chue P, Greenshaw AJ, Agyapong VIO. Enhancing peer support experience for patients discharged from acute psychiatric care: protocol for a randomised controlled pilot trial. BMJ Open. 2018 Aug 17;8(8):e022433. doi: 10.1136/bmjopen-2018-022433. PMID 30121611